CLINICAL TRIAL: NCT04755101
Title: Cardio-Neuromodulation in Humans, 3th Study
Brief Title: Efficacy of a Right-sided Ablation of the Anterior Ganglionated Plexus for Neurally Mediated Syncope
Acronym: CardNMH3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imelda Hospital, Bonheiden (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); AZ Sint-Jan AV (Other); Biosense Webster, Inc. (Industry); Trium Clinical Consulting (Industry)
Responsible Party: Principal Investigator, Philippe Debruyne, Cardiologist, head of Electrophysiology and Research Departments, Imelda Hospital, Bonheiden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3222020000229
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Syncope, Neurogenic; Syncope
Keywords: cardioneuroablation; cardio-neuromodulation; ganglionated plexi; right-anterior ganglionated plexus; ablation
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Righ-sided ARGP ablation (Active Comparator): two-thirds of the patients will be randomized to procedural arm A: a diagnostic evaluation followed by cardio-neuromodulation (CardNM) and a pharmacological evaluation
  Interventions: Procedure: EPS, electro-anatomical mapping, ARGP ablation, and pharmacological evaluation.
- Placebo (Sham Comparator): one-third of the patients will be randomized to procedural arm B: a diagnostic evaluation followed by a pharmacological evaluation.
  Interventions: Procedure: EPS, electro-anatomical mapping, and pharmacological evaluation.

INTERVENTIONS:
Procedure: EPS, electro-anatomical mapping, ARGP ablation, and pharmacological evaluation. — EPS and electro-anatomical mapping of the right atrium and the surrounding veins. A target line (TL) is traced at the posteroseptal side of the junction, between the right atrium and superior vena cava, facing the mid and caudal parts of the right superior pulmonary vein antrum on the right heart cavities on a CT image imported into the CARTO system. This map will be carefully merged with the CT image and the TL will be visible. Sequential ablations will be delivered along theTL until the procedure endpoint is reached. Pharmacological evaluation.
  Arms: Righ-sided ARGP ablation
Procedure: EPS, electro-anatomical mapping, and pharmacological evaluation. — EPS and electro-anatomical mapping of the right atrium and the surrounding veins. A target line (TL) is traced at the posteroseptal side of the junction, between the right atrium and superior vena cava, facing the mid and caudal parts of the right superior pulmonary vein antrum on the right heart cavities on a CT image imported into the CARTO system. This map will be carefully merged with the CT image and the TL will be visible. No ablation is performed (sham). Pharmacological evaluation.
  Other Names: EPS, electro-anatomical mapping, no ablation, and pharmacological evaluation.
  Arms: Placebo

SUMMARY:
The third study on CardNM (CardNMH3 study) is a multicenter, double-blind, randomized trial with a sham control group investigating the efficacy and safety of a computed tomography (CT)-guided, right-sided ablation of the anterior ganglionated plexus to prevent recurrence of syncope in patients with neurally mediated syncope (NMS).

The primary goal of the study is to determine whether a CT-guided, right-sided ablation of the anterior ganglionated plexus safely reduces the risk of recurrent episodes of syncope in patients with a history of recurrent NMS.

Two-third of the patients will be randomized to the active arm and one-third to the control arm (sham).

The study procedure is described in the 'detailed description' and 'intervention description'.

Syncope burden, syncope occurrence and quality of life will be assessed by questionnaires at baseline and at 1, 3, 6 and 12 months. A 24-h rhythm registration will be performed at baseline and at 1-, 3- and 6-month follow-up to investigate the influence of the intervention on heart rate.

The effect of CardNM on blood pressure and on chronotropic sinus node function will be evaluated in 2 additional substudies. Patients enrolled in the blood-pressure substudy will undergo a 24-h blood pressure monitoring at baseline and at 1, 3 and 6 months. Participants in the sinus node competence substudy will undergo a bicycle exercise test at baseline and at 1, 3 and 6 months.

Investigators aim to achieve complete follow-up for 110 patients who meet the study enrollment criteria. If syncope-free survival (primary endpoint) is significantly different between the 2 arms after the enrollment of fewer than 110 patients (minimum 55 patients), enrollment into the trial will be prematurely stopped. The study may also be terminated prematurely if safety concerns occur.

DETAILED DESCRIPTION:
The efficacy of therapeutic strategies mentioned in the guidelines for patients with neurally mediated syncope (NMS) is limited. The first clinical study on cardiac denervation in humans was published in 2005. Derived from this first method, different approaches to cardioneuroablation (CNA) to treat NMS have been published. Such ablations are complex, bi-atrial, and extensive. Cardio-neuromodulation (CardNM) is a less extensive and right-sided approach to CNA, based on a tailored vagolysis of the sinoatrial node through partial ablation of the anterior right-ganglionated plexus. Evidence from a single-center, non-randomized, unblinded trial showed that CardNM was associated with a reduction in syncope burden exceeding 90%.

This third study on CardNM (CardNMH3 study) is a multicenter, double-blind, randomized trial with a sham control group investigating the efficacy and safety of a computed tomography (CT)-guided, right-sided ablation of the anterior ganglionated plexus to prevent recurrence of syncope in patients with neurally mediated syncope.

The primary goal of the study is to determine whether a CT-guided, right-sided ablation of the anterior ganglionated plexus safely reduces the risk of recurrent episodes of syncope in patients with a history of recurrent NMS.

Two-thirds of the patients will be randomized to the active arm and one-third to the control arm (sham).

In all patients, the endocardial site to potentially target during ablation will be annotated before the procedure by a target line (TL) on a computed tomographic image of the heart imported into the CARTO system (Biosense Webster, Diamond Bar, CA), as detailed in the 'intervention description'.

The study procedure will be performed under general anesthesia according to a standardized protocol. In all patients, a diagnostic electrophysiology study (EPS) and electroanatomical mapping of the right atrium and the surrounding veins will be performed first. This image will be merged with the CT image and the TL will be visible. Randomization will be performed electronically at this stage of the procedure.

In patients assigned to the active arm, the TL will be targeted by ablation as detailed in the intervention description'.

The ablation procedure is considered complete when one of the following conditions is fulfilled:

1. 10 radiofrequency applications have been delivered;
2. After 5 radiofrequency applications, the P-P interval is <70% of the baseline procedural P-P interval and remains >550 ms 5 min after the last radiofrequency application;
3. ≥5 radiofrequency applications have been delivered and the operator estimates that no additional P-P interval shortening will be obtained by additional radiofrequency applications;
4. 3 radiofrequency applications have been delivered and the P-P interval is <550 ms after the last radiofrequency application and remains stable after 5 min of waiting.

In all patients, a pharmacological evaluation and new diagnostic EPS will be performed to further evaluate the sinus node and atrioventricular nodal intrinsic activity at the end of the procedure, either after the diagnostic part of the procedure in the sham group or after the ablation in the active arm.

Syncope burden, syncope occurrence and quality of life will be assessed by questionnaires completed at baseline and at 1, 3, 6 and 12 months. A 24-h rhythm registration will be performed at baseline and at 1-, 3- and 6-month follow-up to investigate the influence of the intervention on heart rate.

The effect of CardNM on blood pressure and on chronotropic sinus node function will be evaluated in 2 additional substudies. Patients enrolled in the blood-pressure substudy will undergo a 24-h blood pressure monitoring at baseline and at 1, 3 and 6 months. Participants in the sinus node competence substudy will undergo a bicycle exercise test at baseline and at 1, 3 and 6 months.

Investigators aim to achieve complete follow-up for 110 patients who meet the study enrollment criteria. If the syncope-free survival, the primary endpoint of the study, is significantly different between the 2 arms after the enrollment of fewer than 110 patients (minimum 55 patients), enrollment into the trial will be prematurely stopped. The study may also be terminated prematurely if safety concerns occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be in sinus rhythm and have ≥3 syncopes during the last 18 months* and a previous positive tilt table test (TTT) with a cardioinhibitory or mixed response (VASIS I, IIA or IIB classification).

  * syncopes occurring during TTT are not taken into account
* Patients have a 'preserved cholinergic SN reserve', defined as ≥20% sinus heart rate increment during a pharmacological test with atropine.

Exclusion Criteria:

* <14 years age
* Any unstable medical condition, life expectancy <12 months
* Inability to provide consent or undergo follow-up
* Syncope due to a non-cardiac disease or due to an advanced neuropathy
* Moderate to severe valvular or subvalvular aortic stenosis or mitral stenosis
* Overt heart failure or left ventricular ejection fraction <45%
* Current pregnancy
* Chronotropic negative medications unless judged mandatory
* 4 g amiodarone intake during the 2 months preceding enrollment
* Alternating RBBB and LBBB, HV interval >70 ms
* LBBB, bifascicular block (RBBB + LAHB, RBBB + LPHB)
* PR interval permanently >240 ms
* Pacemaker or automated implantable cardioverter defibrillator device
* Permanent AF, PAF or electrical cardioversion during the last 6 months
* Channelopathy
* Tilt table test with VASIS III response or with VASIS II response and AV-Block

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Syncope free survival | From date of randomization until the date of first syncope recurrence, assessed up to 12-month follow-up.
  The primary efficacy endpoint is the number of days elapsed from study procedure to first syncope recurrence or to study close-out.

SECONDARY OUTCOMES:
Syncope burden | 1-, 3-, 6- and 12-month follow-up.
  Corrected cumulative number of syncope episodes
Number of beats with prespecified P-P intervals | 1-, 3- and 6-month follow-up.
  Mean number of beats with prespecified P-P intervals over 24-h
Heart rate variability | 1-, 3- and 6-month follow-up.
  Standard deviation of the average NN (SDNN)
Quality of life scale based on the questionnaire 'Impact of Syncope on Quality of Life (ISQL) | 1-, 3-, 6- and 12-month follow-up.
  Comparison of scores; higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Debruyne, MD, Principal Investigator — Imeldaziekenhuis
Locations (3):
- Belgium (3):
  - Imeldaziekenhuis, Bonheiden
  - Algemeen Ziekenhuis Sint Jan, Bruges
  - Universitair Ziekenhuis Gasthuisberg, Leuven

IPD SHARING:
Plan to Share IPD: No